CLINICAL TRIAL: NCT06895915
Title: Accuracy of Immediate Implant Placement Using Robotic System Versus Dynamic Navigation System in Anterior Maxillae: a Random Controlled Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, shichong Qiao, Research Fellow, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH9H-2024-T306-2
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Tooth Diseases
Keywords: immediate implant placement; dynamic navigation; robotic surgery
MeSH Terms: conditions — Tooth Diseases | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic Surgery (Experimental): Immediate implant placement assisted by robotic surgery
  Interventions: Procedure: dynamic navigation surgery
- Dynamic navigation (Sham Comparator): Immediate implant placement assisted by dynamic navigation
  Interventions: Procedure: robotic surgery

INTERVENTIONS:
Procedure: dynamic navigation surgery — immediate implant placement assisted by dynamic navigation
  Arms: Robotic Surgery
Procedure: robotic surgery — immediate implant placement assisted by robotic surgery
  Arms: Dynamic navigation

SUMMARY:
Prosthetic-driven immediate implant placement for optimal aesthetic restoration has been increasing in demand during the last decades but requires higher accuracy. Dynamic navigation has been reported better implant positioning in immediate implant placement compared to free hand procedure. On the basis of dynamic navigation, robotic system uses the robotic arm to replace the manual process of implant bed preparation and implant placement, therefore improving the accuracy of implant placement theoretically. The goal of this randomized controlled trial is to compare the positional implant accuracy, the surgical time, and patient satisfaction between dynamic navigation and robotic assisted immediate implant placement in maxillae. Subjects will be randomized to either group based on the allocation. The accuracy of placement will be assessed evaluating the difference between the planned and the actual position using a follow-up CBCT scan taken at the end of the surgery. Subjects will be followed up for one year to assess both patient reported and professional outcomes.

DETAILED DESCRIPTION:
Prosthetic-driven immediate implant placement for optimal aesthetic restoration has been increasing in demand during the last decades but requires higher accuracy. Dynamic navigation has been reported better implant positioning in immediate implant placement compared to free hand procedure. However, dynamic navigation faces the following deficiencies in immediate implant placement. Firstly, it has a steep learning curve. Secondly, the rigid palatal bone wall of the socket will force the direction of drill deviating buccally. On the basis of dynamic navigation, robotic system uses the robotic arm to replace the manual process of implant bed preparation and implant placement, therefore improving the accuracy of implant placement theoretically. The goal of this randomized controlled trial is to compare the positional implant accuracy, the surgical time, and patient satisfaction between dynamic navigation and robotic assisted immediate implant placement in maxillae. Subjects will be randomized to either treatment modalities based on the plan. The accuracy of placement will be assessed evaluating the difference between the planned and the actual position using a follow-up scan taken at the end of the surgery. Subjects will be followed up for one year to assess the professional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* a. ≥18 years old and in good health; b. One or more maxillary incisors that cannot be retained due to non-periodontitis; c. The buccal bone plate is complete; d. No acute infection; e. The extraction socket have at least 3-5 mm apical bone.

Exclusion Criteria:

* a. General contraindications of oral implant surgery (such as immunodeficiency, long-term use of corticosteroids); b. Treatments or diseases that may affect bone tissue metabolism (for example, taking bisphosphonates or receiving local radiotherapy); c. Periodontitis history or uncontrolled periodontitis. Bleeding of probing (BOP) positive site ≥ 10%, or probing depth (PD) ≥ 4mm; d. Heavy smokers or previous heavy smoking history (quit smoking time <5 years or> 20 cigarettes per day); e. Refuse to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Implant positional accuracy | immediately after surgery
  Implant accuracy will be measured as discrepancy between the digital plan and the actual position of the implant.

SECONDARY OUTCOMES:
Surgery time | intraoperative
  Time needed for surgery procedure will be recorded from anaesthesia to connection of cover screw/healing abutment.
Pain perception | Immediately after surgery
  Patient pain perception during surgery will be recorded using visual analogue scale (VAS with range from 0 to 10 with 10 being the highest possible pain experience).
Pain perception | 7 days after surgery
  Patient pain perception after surgery will be recorded using visual analogue scale (VAS with range from 0 to 10 with 10 being the highest possible pain experience).
Surgeon preference | Immediately after surgery
  Assessed using a visual analogue scale (VAS, 100 mm, with 0=least desirable option and 100 = most desirable option.
Soft tissue changes | immediately after crown delivery
  Assessed by midfacial recession, mesial and distal papillary recession.

IPD SHARING:
Plan to Share IPD: Undecided